CLINICAL TRIAL: NCT05763251
Title: Short Course Versus Standard Course Antifungal Therapy for Uncomplicated Candidemia in Children and Adolescents: A Multi-Center Randomized Controlled Trial
Brief Title: Comparison of Uncomplicated Candidemia Therapy Duration in Children
Acronym: COUNT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: Westat (Other); St. Jude Children's Research Hospital (Other); George Washington University (Other); Children's Hospital of Philadelphia (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-020057; 1R01AI170385-01 (NIH)
Record Dates: First submitted 2023-02-23; First posted 2023-03-10 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-09

CONDITIONS: Invasive Candidiasis
MeSH Terms: conditions — Candidiasis, Invasive | interventions — Duration of Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Short-course therapy (Experimental): pediatric patients with uncomplicated candidemia who have already received 7 days of primary systemic antifungal therapy will receive no additional antifungal therapy
  Interventions: Other: therapy duration
- Standard-course therapy (No Intervention): pediatric patients with uncomplicated candidemia who have already received 7 days of primary systemic antifungal therapy will receive 7 additional days of systemic antifungal therapy

INTERVENTIONS:
Other: therapy duration — the standard-course arm will receive 14 days total of antifungal therapy and the short-course arm will only receive 7 days of therapy
  Arms: Short-course therapy

SUMMARY:
The goal of this clinical trial is to compare antifungal therapy duration in pediatric uncomplicated candidemia. The specific aims are:

* Compare the desirability of outcome ranking in children with uncomplicated candidemia randomized to 7 additional days of antifungal therapy (standard-course) versus no additional antifungal therapy (short-course) after already receiving 7 days of echinocandin therapy.
* Compare the 14-day desirability of outcome measure for subjects with a negative and those with a positive T2Candida® biomarker at day 7 of therapy within randomized groups.

Participants meeting eligibility criteria will be approached and consented between day 5 and 7 of primary systemic antifungal therapy. On day 7 of primary systemic antifungal therapy, inclusion and exclusion criteria will again be reviewed for consented patients and those still eligible will be randomized 1:1 to the two study arms. Researchers will compare no additional antifungal therapy (short-course) versus 7 additional days of systemic antifungal therapy (standard-course) in pediatric patients with uncomplicated candidemia who have already received 7 days of primary systemic antifungal therapy to see if shorter durations are as effective as longer durations in treating uncomplicated candidemia.

DETAILED DESCRIPTION:
The primary objective of this study will be addressed with a multi-center open label randomized controlled trial designed to compare no additional antifungal therapy (short-course) versus 7 additional days of systemic antifungal therapy (standard-course) in pediatric patients with uncomplicated candidemia who have already received 7 days of primary systemic antifungal therapy. The secondary objective of this study is an embedded observational biomarker study. This objective will determine if the novel T2Candida® biomarker performed at the time of randomization (i.e. Day 7 of systemic antifungal therapy) will be associated with patient outcomes assessed at Day 14. The results of the T2Candida® biomarker will not be available in real-time and thus will not impact the primary study objective. Eligible patients will be any hospitalized patient at a participating center with uncomplicated candidemia that is older than 120 days and <18 years of age at time of candidemia onset. Patients need to receive an echinocandin as their primary antifungal therapy for at least three days and continue systemic antifungal therapy (either with an echinocandin or step-down to an azole) for a total of 7 days from their first negative blood culture and have no evidence of metastatic foci of candidemia at the time of randomization. Patients with neutropenia or anticipated to have neutropenia during the study follow-up window will not be eligible. Patients can only be enrolled to the study once. This study population will serve as the source cohort for both study objectives. Patients will be randomized 1:1 to one of two study arms, short-course therapy or standard-course therapy. Patients will be followed for 21 days from the day of randomization (Day 7 to Day 28) to capture primary and secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 120 days and < 18 years at the time of positive blood culture at any participating site;
2. Candidemia with at least one positive blood culture for any Candida spp;
3. Receiving/received an echinocandin (caspofungin, micafungin or anidulafungin) as primary antifungal therapy for candidemia for at least 2 days from day of first negative culture with continuation of uninterrupted systemic antifungal therapy at the time of enrollment);
4. Sustained clearance of Candida spp. from repeat blood culture(s) obtained on or before day of randomization;
5. Partial or complete clinical response, as defined by published guidelines, on or before day of randomization;
6. No evidence of metastatic foci of infection at the time of randomization, as documented by a negative abdominal ultrasound or abdominal CT scan of the liver, spleen, and kidneys and negative ophthalmologic examination.

Exclusion Criteria:

1. Already receiving antifungal therapy for a previously diagnosed systemic invasive fungal disease;
2. Neutropenic (absolute neutrophil count < 500 cells/μl) at the time of enrollment or anticipated to be neutropenic in the week following randomization;
3. Have an underlying condition that requires them to be on antifungal prophylaxis when not receiving directed therapy for an invasive fungal disease;
4. Previous enrollment in this trial.
5. Females of childbearing age with a current pregnancy diagnosis or without a negative pregnancy test for their current admission
6. A documented DNR order
7. Have an implantable cardiac device (e.g., ventricular assist device, pacemaker)

Ages: 120 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Compare the desirability of outcome ranking (DOOR) in short-course vs standard-course arm | The measures assigned on Day 14 will inform the primary analysis for the primary objective
  The primary analysis for the primary objective will compare the DOOR distributions at 7 days from randomization (i.e., outcome assessment on Day 14 from first negative blood culture) between subjects from the two study groups, based on randomized treatment assignments, in accordance with the intention-to-treat principle. The primary analysis will use the DOORs assigned on this day to assess which therapy course is better, short-course or standard-course.

SECONDARY OUTCOMES:
Compare the DOOR for subjects with a negative vs positive T2 Candida® biomarker at day 7 | The DOOR measure on Day 14 will be used for the primary analysis for the secondary objective.
  The results of the Day 7 T2Candida® biomarker (i.e. detected versus not detected) and the randomization group (i.e. short-course versus standard-course) will allow for the following four subsets of patients: 1. Patient is randomized to short-course group and has a not-detected result for the T2Candida® biomarker at time of randomization; 2. patient is randomized to short-course group and has a detected T2Candida® biomarker at time of randomization; 3. patient is randomized to standard-course group and has a not-detected result for the T2Candida® biomarker at time of randomization; 4. patient is randomized to standard-course group and has a detected T2Candida® biomarker at time of randomization. This analysis will compare the DOOR categories between the first two groups (i.e. short-course and not-detected versus short-course and detected) and then be repeated for the second two groups (i.e. standard-course and not detected versus standard-course and detected).

CONTACTS AND LOCATIONS:
Overall Officials: Brian Fisher, DO, Principal Investigator — Children's Hospital of Philadelphia; William J Steinbach, MD, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (17):
- United States (17):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Orange County, Orange, California
  - Yale New Haven Children's Hospital, New Haven, Connecticut
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Comer Children's Hospital, Chicago, Illinois
  - Riley Children's Hospital, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Weill Cornell Medical College, New York, New York
  - Duke Children's Hospital, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Dell Children's Medical Center, Austin, Texas
  - Primary Children's Hospital, Salt Lake City, Utah